CLINICAL TRIAL: NCT07282847
Title: A Single-Arm, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability and Efficacy of a Single Intravenous Infusion of AB-1009 in Adult Participants With Late Onset Pompe Disease (LOPD)
Brief Title: A Study to Evaluate Safety, Tolerability, and Efficacy of AB-1009 Gene Therapy (GAA Gene) in Adult Participants With Late Onset Pompe Disease (PROGRESS-GT LOPD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASK-POM9-CS101
Record Dates: First submitted 2025-11-26; First posted 2025-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease (Late-onset); Pompe Disease Late-Onset; LOPD
Keywords: Pompe Disease; Glycogen Storage Disease; Lysosomal Storage Diseases; Acid Maltase Deficiency; Acid Maltase Deficiency Disease; Gene Therapy; AB-1009; Neuromuscular Disease; LOPD; Acid-Alpha Glucoside (GAA); GAA gene; Adeno-Associated Virus (AAV); Late-Onset Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II; Glycogen Storage Disease; Lysosomal Storage Diseases; Neuromuscular Diseases | interventions — alpha-Glucosidases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 1.0E13 vg/kg
  Interventions: Genetic: AB-1009 (GAA Gene)
- Cohort 2 (Experimental): 1.5E13 vg/kg
  Interventions: Genetic: AB-1009 (GAA Gene)

INTERVENTIONS:
Genetic: AB-1009 (GAA Gene) — A single intravenous infusion of AB-1009

SUMMARY:
This is a single-arm, open-label, dose-escalation study to evaluate the safety, tolerability and efficacy of a single intravenous infusion of AB-1009 in adult participants with late-onset Pompe disease (LOPD).

DETAILED DESCRIPTION:
This is an open-label study, up to 12 participants will receive a single IV infusion of AB-1009. Participants will be assigned to either cohort 1 (1.0E13 vg/kg) or Cohort 2 (1.5E13 vg/kg) based on enrollment in the study.

Study duration will include a screening period of up to 75 days, primary observation of 52 weeks, and a long-term follow-up period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age at the time of signing the informed consent form.
2. Confirmed GAA enzyme deficiency from any tissue source and/or confirmed biallelic GAA gene mutations.
3. Undergone enzyme replacement treatment (ERT) (either alglucosidase alfa (Lumizyme®) or avalglucosidase alfa-ngpt (Nexviazyme®)), for at least 6 months (at least 10 infusions) before signing the initial informed consent form. During the screening process, participants need to remain on their current ERT until close to dosing;
4. FVC in the upright position ≥30% and ≤80% of predicted;
5. Capable of walking at least 100 meters in the 6MWT (use of a cane, quad cane, or standard walker is permitted);
6. Contraceptive/barrier use by men and women requirements as per protocol.
7. Capable of giving informed consent and able to understand and comply with all study procedures.

Exclusion Criteria:

1. Severe cardiomyopathy, defined as left ventricular ejection fraction (LVEF) <40% or New York Heart Association (NYHA) functional class 3 or above;
2. Require invasive mechanical ventilation, or rely on noninvasive ventilation during the day;
3. Intolerance to ERT or investigator-assessed intolerance to ERT, prior experience of serious ERT-related infusion-associated reactions (IARs);
4. Have known intrinsic liver diseases, including hepatitis, HIV-related liver disease, prior diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy, severe fatty liver, cirrhosis or liver fibrosis ≥stage 2, ultrasound-identified liver neoplasms, or laboratory tests suggesting elevated alpha-fetoprotein. Patients with liver function tests including ALT or AST >3× upper limit of normal (ULN) or any total bilirubin above ULN during screening will also be excluded;
5. Prior or ongoing medical condition(s), physical finding(s), assessment findings, or laboratory abnormality that, in the investigator's opinion, would impact participant's safety and compliance with the study procedures.
6. Have received gene therapy prior to screening;
7. Have received any systemic immunosuppressants (except inhalation or topical use) other than glucocorticoids or investigator-recommended immunosuppressants 30 days prior to screening through completion of screening, and/or known intolerance to immunosuppressants such as glucocorticoids;
8. Use of investigational drugs or drugs that could affect this study as evaluated by the investigator within 30 days prior to screening through completion of Week 52 or within 5 half-lives of the investigational drug (whichever is longer);
9. Have received any vaccine within 30 days prior to dosing;
10. Other conditions that make the participant not eligible for the study according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Day 1 (Dosing) to Week 52 (the end of the primary observation period)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, Irvine (UCI), Irvine, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - NYU Langone, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University of Texas Southwest Medical Center, Dallas, Texas
  - Virginia Commonwealth University (VCU), Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No